CLINICAL TRIAL: NCT04997434
Title: Impact of Modern Art Therapy on Patients' Anxiety and Pain During the Waiting Time in an Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier Hugli (Other)
Responsible Party: Sponsor-Investigator, Olivier Hugli, Principal investigator, promoter, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-01344
Record Dates: First submitted 2021-07-19; First posted 2021-08-09 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Anxiety Acute; Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After 5-10 minute interview with the patient to define his or her tastes and contraindications to certain techniques. The patient will have 15 to 20 minutes to carry out an artistic activity, accompanied by the art therapist according to his/her needs. During the activity, verbal exchanges will continue. After the session, 5 minutes will be devoted to the patient's self-evaluation of the past moment, of his level of anxiety, of the intensity of his pain and of his feelings in relation to his passage in the Emergency Department and the art therapy session.
  Interventions: Behavioral: Art-therapy in the emergency department
- Control (No Intervention): The questionnaires and VAS will be offered to the control group at the beginning of the wait, then after 30 minutes of waiting under usual conditions.

INTERVENTIONS:
Behavioral: Art-therapy in the emergency department — The intervention will begin with a 5-10 minute interview with the patient to define his or her tastes and contraindications to certain techniques. Since the art-therapeutic intervention that will be proposed seeks to generate pleasant feelings, it will be important to rely on the patient's tastes. At the end of the interview, modern art therapy will be presented to the patient and several artistic activities will be proposed (origami, drawing, creative writing).
  Once the activity has been chosen, the patient will have 15 to 20 minutes to carry it out, accompanied by the art therapist according to his/her needs. During the activity, verbal exchanges will continue. After the 15 to 20 minutes of the session, 5 minutes will be devoted to the patient's self-evaluation of the past moment, of his level of anxiety, of the intensity of his pain and of his feelings in relation to his passage in the Emergency Department and the art therapy session.
  Arms: Intervention

SUMMARY:
The primary objective of this study is to investigate whether, during a waiting period in an emergency department, the patient's participation in a modern art therapy session decreases the patient's level of anxiety and pain.

As a secondary objective, this study aims to explore whether participation in a modern art therapy session is perceived positively by the patient. This objective will be assessed by both patient self-report and art therapist heteroreport.

In this work, the investigators will therefore seek to demonstrate the potential positive impact of modern art therapy conducted during times of waiting for examination or results.

DETAILED DESCRIPTION:
After reviewing the patients' medical records in the emergency department, and verifying the inclusion and exclusion criteria with the caregivers in charge of the case, the investigators will introduce themselves to the patients and offer them to participate in the study. The investigators will explain to the patients that their emergency department experience involves waiting time and that they are eligible for this study aimed at improving the well-being of emergency department patients during waiting time. Patients will be informed that the study aims to investigate the distracting effect of a modern art therapy session. If the patients ask about the modalities of the session, the investigators will answer that it will consist of an artistic production in accordance with their tastes and abilities, defined with the art therapist or a discussion with the research nurse about art therapy and its place in an emergency department and that they will be randomly assigned to one of the two groups.

At this stage, only oral consent will be obtained. After verifying that all inclusion criteria are met, that none of the exclusion criteria are applicable, and obtaining oral consent, each patient will be randomized 1:1 between the two study arms using the randomization module in the RedCap® software. The investigator in charge of data collection will collect some additional data in a standardized way by following the case report form.

The art therapist will then be able to intervene with the patient if the latter is part of the group participating in an art therapy session. A five- to ten-minute interview with the patient will allow the art therapist to get to know the patient and to learn more about his or her tastes and any contraindications the patient may have to certain techniques. This interview will begin with a discussion of the patient's general condition, both physical (pain, injury) and mental (mood), with the goal of assessing preserved and mobilizable abilities as well as affected and non-mobilizable mechanisms. The patient's tastes (artistic or other) will also be briefly questioned. Since the art-therapeutic intervention that will be proposed seeks to generate pleasant feelings, it will be important to rely on the patient's tastes. It is the patient's tastes and choices that will guide the decision of the dominant artistic elements, in order to maximize the pleasure taken in the activity and the distracting effect of the proposal. At the end of the interview, modern art therapy will be presented to the patient and several artistic activities will be proposed:

* Origami: paper folding activity requiring good fine motor skills, possible if the patient can fully use his/her hands. Requires a flat surface to put the paper on.
* Drawing: with dry techniques that will be disinfected after each use. It could be a drawing of invention, a comic strip to complete, an extension of a photo by a drawing...
* Writing: with markers or pens to allow for quick drying and avoid smearing. Creative writing games working on the imagination can be proposed.

All paper elements intended to be contemplated (models or works of art) will be wrapped in plastic to allow disinfection between each use.

Once the activity has been chosen, the patient will have 15 to 20 minutes to carry it out, accompanied by the art therapist according to his/her needs (explanations, gestural and technical support, partial or total realization by the art therapist under the patient's orders...). During the activity, verbal exchanges will continue. After the 15 to 20 minutes of the session, 5 minutes will be devoted to the patient's self-evaluation of the past moment, of his level of anxiety, of the intensity of his pain and of his feelings in relation to his passage in the Emergency Department and the art therapy session. The question will then be raised as to what will happen to the production, which will either be discarded or given to the patient to take with him/her.

The materials used for this study are common plastic arts materials (pencils, markers, paper) that are non-toxic and non-dirty. Reproductions of artworks in the form of postcards may also be shown to the patients.

For the control group without art therapy, the patient will be left in the usual waiting conditions for 20 to 30 minutes. After this waiting time, the patient will be asked to self-assess his or her level of anxiety, pain intensity and feelings about his or her visit to the emergency department.

Once all the data has been collected, a complete information sheet and a consent form will be given to the patient. Additional explanations can be given upon request. Patients will have a minimum of 15 minutes to sign the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patient whose management requires waiting for a procedure, an examination or results
* Patient whose pain is evaluated at least 3/10 by a VAS on arrival in the emergency room.

Exclusion Criteria:

* Clinically unstable patients (i.e., admitted to the intensive care unit or deemed unstable by the physician or nurse responsible for the patient)
* Patient incapable of judgement or with whom it is difficult to communicate
* Altered mental status (e.g. cognitive impairment, mental retardation, acute confusional state, acute psychosis)
* Intoxication
* Alcohol abuse
* Patient unable to communicate in French at a level sufficient to give informed consent and answer questions related to their anxiety and pain
* Patient unable to understand the use of VAS scales
* Patient incarcerated
* Patient transferred from another hospital
* Patient who has participated in this study at a previous visit
* Patient with chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Anxiety self-assessment | Up to 4 hours (from admission in the departement to end of session)
  The primary outcomes of this study will be patients' self-assessment of their anxiety status using a visual analog scale and a validated questionnaire This measurement will be taken before and after an art therapy session during their waiting time in the emergency department.
Anxiety self-assessment | Up to 4 hours (from admission in the departement to end of session)
  The primary outcomes of this study will be patients' self-assessment of their anxiety status using the State-Trait Anxiety Inventory. This measurement will be taken before and after an art therapy session during their waiting time in the emergency department.
Pain self- assessment | Up to 4 hours (from admission in the departement to end of session)
  The primary outcomes of this study will be patients' self-assessment of their pain intensity using a visual analog scale. This measurement will be taken before and after an art therapy session during their waiting time in the emergency department.
Anxiety assessment | 20 minutes (during the session)
  The art therapist will also assess the patient's anxiety during the session using items that allow the recording of observable phenomena on a scale from 1 to 5, 1 beeing the worse outcome, 5 the best.
Pain assessment | 20 minutes (during the session)
  The art therapist will also assess the patient's pain during the session using items that allow the recording of observable phenomena on a scale from 1 to 5, 1 beeing the worse outcome, 5 the best.

SECONDARY OUTCOMES:
Pleasure self-assessment | 1 minute (end of session)
  The secondary results of this study will be the patient's self-evaluation by visual analog scale of the pleasure felt during the activity. 1 will be the worse outcome, 10 the best.
Feeling towards the passage in the emergency department | 1 minute (end of session)
  Questions will be asked to the patient regarding how he feels about his passage in the emergency department. The possible answers will be "poor", "fair", "good", "excellent". They will be converted in numbers from 1 to 4, 4 (excellent) being the best outcome.
Quality of realization self-assessment | 1 minute (end of session)
  The secondary results of this study will be the patient's self-evaluation by visual analog scale of the quality of its realization.1 will be the worse outcome, 10 the best.
Aesthetic pleasure self-assessment | 1 min (end of session)
  The secondary results of this study will be the patient's self-evaluation by visual analog scale of the aesthetic pleasure felt in front of their realization. 1 will be the worse outcome, 10 the best.
Pleasure towards the activity self-self assessment | 1 min (end of session)
  The secondary results of this study will be the patient's self-evaluation by visual analog scale of the pleasure expressed towards the activity. 1 will be the worse outcome, 10 the best.
Engagement of the patient in the activity assessment | 20 minutes (during the session)
  The engagement of the patient in the activity during the session will also be evaluated by the art-therapist using items that allow the recording of observable phenomena on a scale from 1 to 5, 1 beeing the worse outcome, 5 the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No